CLINICAL TRIAL: NCT05553158
Title: Study to Investigate the Influence of Compression Treatment in Patients With Pelvic Congestion Syndrome (PCS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Whiteley Clinic (Other)
Collaborators: Bauerfeind (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TWC-AC-2021-03
Record Dates: First submitted 2021-09-01; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Pelvic Congestive Syndrome

STUDY DESIGN:
Intervention Model Description: There are two arms in this study: control arm and interventional arm. Participants in the control arm will have pelvic vein embolization and participants in the interventional arm will have compression therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pelvic Vein Embolization (PVE) (Active Comparator): Patients will have their pelvic veins embolized in accordance with their personalised treatment plan, based on their trans-vaginal ultrasound scan. These patients form the control group.
  Interventions: Device: Embolization coils
- Compression Therapy (Experimental): Patients will wear compression pants (with leg compression if patients also have symptomatic leg varicose veins).
  Interventions: Device: Compression pants

INTERVENTIONS:
Device: Compression pants — Similar to compression stockings for the legs which are designed to apply pressure to improve venous return in the legs, compression pants have been designed to apply pressure to pelvic veins to improve the symptoms of Pelvic Congestion Syndrome.
  Arms: Compression Therapy
Device: Embolization coils — Embolization coils are used to block the veins they are positioned in. This is a standard treatment offered to patients at The Whiteley Clinic.
  Arms: Pelvic Vein Embolization (PVE)

SUMMARY:
Pelvic vein embolization (PVE) is the current treatment procedure used to treat women with Pelvic Congestion Syndrome (PCS). This treatment is not widely available, and many women when diagnosed with PCS cannot afford treatment.

The purpose of this study is to assess whether compression therapy is an effective alternative treatment to PVE for women who are unwilling or unable to undergo treatment by PVE. Compression therapy would provide a cost-effective alternative to coil embolization.

DETAILED DESCRIPTION:
Women that book a consultation and have a trans-vaginal ultrasound scan at The Whiteley Clinic which confirms a diagnosis of Pelvic Congestion Syndrome (PCS) will be informed about the opportunity to participate in this study by their consultant (provided they also fulfil the inclusion/exclusion criteria). Potential participants will be given an information sheet and time to consider the study before giving written informed consent.

These women will be given a personalised pelvic vein embolization (PVE) treatment plan. Women that opt for PVE will form the control group for this study. Women that do not wish to have PVE and opt compression therapy will form the intervention group for this study. Alternatively, women may wish to not have any treatment and will not be enrolled in the study.

Each patient will be directly involved in the study for three months (Month 1, Month 2, Month 3). A quality of life and symptom questionnaire will be completed by all patients at the start of Month 1 (baseline), at the end of Month 2 (1-month post PVE or compression therapy), and at the end of Month 3.

ELIGIBILITY:
Inclusion Criteria

* Females aged 18 - 65 years
* Having one or more symptoms of PCS
* Symptoms: Aching / dragging in pelvis on sitting and/or standing, aching/tender /painful vulval varicose veins, irritable bowel, irritable bladder, deep dyspareunia, low back pain, hip pain with no or very mild changes on hip x-ray.
* Able to understand study and give written consent.
* Able to have trans-vaginal ultrasound scan and attend for follow-up.

Exclusion Criteria

* Under 18 years of age or over 65 years of age
* Currently pregnant, actively trying to get pregnant, planning pregnancy within next 12 months or within 3 months of child-birth
* Current symptoms due to diagnosed gynaecological conditions
* Current or previous malignancy
* Unable or refuse to consent to trans-vaginal ultrasound scan or any other aspect of the study
* Previous abdominal or pelvic surgery (excluding diagnostic laparoscopy)
* Previous embolization of pelvic veins
* Previous deep vein thrombosis, pelvic embolisation, venous intervention in abdomen or pelvis (stent, filter)
* Any vascular malformation of the pelvis or the legs apart from that diagnosed as venous reflux disease.
* Any medical condition likely to cause death or serious ill health within the next five years.
* Any deep venous obstruction or reflux on duplex ultrasound.
* Unable to wear compression garments on lower abdomen / pelvis
* Unable to wear leg compression garments

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Quality of Life and Symptoms at one month post-treatment and at two months post-treatment | Baseline (start of month 0), 1 month post-treatment (end of Month 2) and two months post-treatment (end of month 3)
  Patients will fill out a quality of life and symptoms questionnaire at the start of the study (baseline (month 0)). Patients will then undergo treatment after one month. A quality of life and symptoms questionnaire will then be filled out again one month after treatment (end of month 2), and again a month later (end of month 3). This questionnaire uses visual analogue scales to quantify quality of life and the severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Whiteley, MS FRCS(Gen) MBBS, Principal Investigator — The Whiteley Clinic
Locations (1):
- The Whiteley Clinic, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No